CLINICAL TRIAL: NCT04558983
Title: A Natural History Study to Evaluate Functional and Anatomical Progression in Retinitis Pigmentosa
Status: Terminated | Type: Observational
Why Stopped: The study stopped because patients dropped out of the study to participate in the interventional trials. With interventional trials present there is very little interest in participating in a Natural Histoy study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00227603
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retinitis Pigmentosa: Patients with Retinitis Pigmentosa

SUMMARY:
This study will assess the progression of RP as seen on newer modalities including spectral-domain optical coherence (SD-OCT) and macular assessment integrity (MAIA) microperimetry to evaluate disease status. Understanding the natural history of the disease is not only essential to monitoring and comparing patient populations in clinical trials. It is also fundamental in the predevelopment phase in order to optimize the study duration needed to observe a statistically significant outcome. Furthermore, since the progression of RP is usually slow, relying on traditional tests can take an unfeasible length of time to observe any meaningful changes and assess therapeutic efficacy for new drugs. Therefore, the results of this study will be beneficial in establishing reliable endpoints and outcome measures for future clinical trials. Such outcome measures may be able to detect treatment response with more precision. More importantly, investigators may be able to detect changes early enough to prevent irreversible vision loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients diagnosed with Retinitis Pigmentosa
* Ability to provide informed consent
* Ability to authorize use and disclosure of protected health information

Exclusion Criteria:

* Concomitant ocular pathology that limits central macular function, including but not limited to age-related macular degeneration, diabetic retinopathy, and retinal vein occlusion
* If EZ width ≤200µm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Retinitis Pigmentosa
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change in mean macular sensitivity (dB) over time as assessed by microperimetry | Baseline, every six months up to 2 years
  Microperimetry (MAIA) will be used to test whether there is a change in sensitivity (dB) in the macula

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity (BVCA) | Baseline, every six months up to 2 years
  Scoring will be determined by the number of letters gained or lost per month using Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score and visual acuity score together with an overall score range of 0 to 20/20 where 0 is the worst vision and 20/20 is the best.
Change in Ellipsoid Zone (EZ) width | Baseline, every six months up to 2 years
  This will be assessed by spectral domain optical coherence tomography (SD-OCT)
Change in Quality of Life survey metrics | Baseline, every year up to 2 years
  Scoring will be determined by the National Eye Institute's Visual Function Questionnaire (NEI-VFQ-25). It has 25 question elements each with score ranging from 1(excellent) to 6(very poor), therefore a total minimum score of 25 and maximum score 150.
Change in mean retinal sensitivity | Baseline and at 2 years
  Static Octopus Perimetry will be used to test whether there is a change in mean retinal sensitivity over time using its 30-2 program with III target
Correlation between change in visual functional and anatomical measures | Baseline, every six months up to 2 years
  Change in visual function parameters such as Best Corrected Visual acuity (measured using ETDRS and visual acuity scale), mean macular sensitivity (quantified using MAIA microperimetry), mean retinal sensitivity (quantified using static Octopus perimetry) will be correlated to anatomical parameters such as Ellipsoid width (measurement on Optical Coherence Tomography)
Correlation between change in visual functional measures and Quality of Life survey metrics | Baseline, every year up to 2 years
  Change in Quality of Life survey metrics (Scored using National Eye Institute's Visual Function Questionnaire, NEI-VFQ-25) will be compared to visual function parameters such as Best Corrected Visual acuity (measured using ETDRS and visual acuity scale), mean macular sensitivity (quantified using MAIA microperimetry), mean retinal sensitivity (quantified using static Octopus perimetry)

OTHER OUTCOMES:
Correlation between baseline functional and anatomical measures | Baseline, up to 2 years
  Visual function parameters at baseline such as Best Corrected Visual acuity (measured using ETDRS and visual acuity scale), mean macular sensitivity (quantified using MAIA microperimetry), mean retinal sensitivity (quantified using static Octopus perimetry) will be correlated to anatomical parameters at baseline such as Ellipsoid width (measurement on Optical Coherence Tomography)
Correlation between baseline functional measures and Quality of Life survey metrics | Baseline, up to 2 years
  Visual function parameters at baseline such as Best Corrected Visual acuity (measured using ETDRS and visual acuity scale), mean macular sensitivity (quantified using MAIA microperimetry), mean retinal sensitivity (quantified using static Octopus perimetry) will be correlated to baseline Quality of Life survey metrics (Scored using National Eye Institute's Visual Function Questionnaire, NEI-VFQ-25)
Correlation between functional, anatomic and Quality of Life measures | Baseline, up to 2 years
  Visual function parameters such as Best Corrected Visual acuity (measured using ETDRS and visual acuity scale), mean macular sensitivity (quantified using MAIA microperimetry), mean retinal sensitivity (quantified using static Octopus perimetry), anatomical parameters such as Ellipsoid width (measurement on Optical Coherence Tomography) Quality of Life survey metrics (Scored using National Eye Institute's Visual Function Questionnaire, NEI-VFQ-25) will be correlated.
Proportion of eyes with ≥ 5 loci that show ≥ 6 decibels (dB) decline in mean macular sensitivity from baseline | Baseline, every six months up to 2 years
  This will be measured using MAIA microperimetry
Proportion of eyes with ≥ 5 loci that show ≥ 7 decibels (dB) decline in mean retinal sensitivity from baseline | Baseline and at 2 years
  This will be measured by static Octopus perimetry using 30-2 program with III target

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute at Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No